CLINICAL TRIAL: NCT00486733
Title: Prospective Randomized Trial of Standard Wound Care Versus Standard Wound Care Plus Shock Wave Therapy for Traumatic Wounds of the Extremity
Brief Title: Study to Determine if Shock Wave Therapy Applied to Traumatic Wounds of the Extremity Improves Healing Time
Acronym: CWI
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Collaborators: Tissue Regeneration Technologies (Industry)
Responsible Party: Principal Investigator, Alexander Stojadinovic, Director, Combat Wound Initiative Program, Walter Reed National Military Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06-20028
Record Dates: First submitted 2007-06-13; First posted 2007-06-15 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Soft Tissue Injuries
Keywords: extracorporeal shock wave therapy; soft tissue wounds
MeSH Terms: conditions — Soft Tissue Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of Care (No Intervention): Standard of Care Treatment; no study treatment
- Standard of Care plus Study Treatment (Experimental): Standard of Care Treatment plus study treatment
  Interventions: Device: DermaGold

INTERVENTIONS:
Device: DermaGold — The first four follow-up study assessment and data collection points will coincide with scheduled operative interventions on the wound guided by clinical situation and the treating physician's judgment (approximately every 3-4 days). Subsequent follow-up study assessment and data collection points will occur on study days 28 ± 3, 42 ± 3, 60 ± 3, and 90 ± 3.
  Arms: Standard of Care plus Study Treatment

SUMMARY:
The purpose of this study is to determine if adding shock wave therapy to standard-of-care wound treatment for traumatic extremity wounds helps them heal faster.

DETAILED DESCRIPTION:
Timely return of combat wounded to functional lives and duty is imperative. Reliance upon traditional wound management principles is restrictive, and a treatment paradigm aimed at high-energy projectile contaminated wounds suits the requirements of our combat casualty care program. The nature of war wounds makes them unsuitable for conventional, saline-soaked-gauze dressings.

Extra-corporeal-shockwave-therapy (ESWT) has been used successfully for orthopedic soft tissue indications. Pilot studies indicate that ESWT enhances tissue healing through growth-factor release and neovascularization, with favorable safety profile and anti-bacterial effect, particularly in problematic wounds including fracture non-unions, post-traumatic wounds, and burns.

The need to improve the healing and quality-of-life of the combat wounded, the potential of this minimal-risk technology to improve healing of difficult-to-treat orthopedic/soft tissue injury and infection, as well as the combat casualty care experience of surgeons at WRAMC, dovetail uniquely to have our wounded soldiers and medical center play a pivotal role as the fundamental proving ground and primary beneficiary of this technology.

Comparison(s): Standard-of-care wound therapy compared to standard-of-care wound therapy + ESWT for extremity wounds with the aim of conducting a definitive critical analysis of the role of ESWT in improved treatment and outcomes of traumatic soft tissue injuries of the extremity.

ELIGIBILITY:
Inclusion Criteria:

* Patients should be 18 years of age or older, and capable of providing informed consent indicating awareness of the investigational nature of this trial, in keeping with institutional policy.
* Written informed consent must be obtained from each patient prior to entering the study.
* Female patients will not be pregnant. Exclusion of the possibility of pregnancy by HCG testing (urine or serum) or by history (tubal ligation, hysterectomy, or menopause) is required prior to inclusion in the study.
* Patients should be willing to be followed within the military healthcare system, or the participating civilian center during the course of study treatment and follow-up.
* Patients with traumatic wound(s) of the upper and/or lower extremity. The study wound is the wound with the highest Red Cross Wound Classification (RCWC).
* Patients should demonstrate adequacy of limb perfusion by all of the following clinical parameters in the affected extremity to be treated by investigational shock wave therapy: Palpable distal extremity pulse; Absence of compartment syndrome; or Ankle Brachial Index(ABI) ≥ 0.9 or transcutaneous pulse oximetry, tcP02≥20mmHg.
* Patients with non-circumferential, second degree burn wounds of the upper and/or lower extremity.

Exclusion Criteria:

* Patients with current participation in another clinical investigation of a medical device or a drug the requirements of which may preclude complete involvement in this study.
* Women who are pregnant.
* One or more of the following findings in the affected extremity to be treated by investigational shock wave therapy: Ankle Brachial Index < 0.9 or tcP02<20 mmHg; Significant arterial or venous injury requiring surgical intervention; or Lymphedema.
* Subject has another non-superficial wound near the study wound that is less than 3cm from the study wound or that has a RCWC of 3.
* Active or previous (within 60 days prior to the study screening visit) chemotherapy.
* Active or previous (within 60 days prior to the study screening visit) radiation to the affected extremity to be treated by investigational shock wave therapy.
* Physical or mental disability or geographical concerns (residence not within reasonable travel distance) that would hamper compliance with required study visits.
* The Investigator believes that the subject will be unwilling or unable to comply with study protocol requirements, including the shock wave treatment procedure, standard-of-care self-care requirements, and all study-related follow up visit requirements.
* Patients with 1st degree, 3rd degree, or circumferential extremity burns considered for treatment by investigational shock wave therapy.
* History of sickle cell anemia.
* History of infection with Human Immunodeficiency Virus.
* History of immunodeficiency disorders.
* Severe anemia - Hgb < 7 g/dl (males) or < 6.5 (females).
* Deep vein thrombosis within 6 months of study screening visit.
* Chronic renal insufficiency requiring dialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 213 (Estimated)
Dates: Start 2007-04; Primary Completion 2014-10 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Time to complete wound healing. For purposes of this study, the definition of "healed" is wound closure with total epithelialization of the soft tissue defect, confirmed at two consecutive study visits. | 90 days following initial treatment

SECONDARY OUTCOMES:
Total number of study subjects with a final status of "healed" in the ESWT therapy group versus control group. | 90 days following initial treatment
The percentage of the soft tissue wound that has healed at 90 days as assessed by planimetric computerized digital measurement. | 90 days following intitial treatment
The number of shock wave treatments performed. | Within six weeks following initial treatment
For patients who have not achieved healed status at Day 90, the percent of wounds at Day 90 with lesser healing (≤50% epithelialization) versus with greater healing (>50% but < 100% epithelialization) as determined by planimetric CDM. | 90 days following initial treatment
Results of quantitative wound bacterial cultures (wounds with a quantitative wound bacterial count greater than 105 per gram of tissue will be defined as an "infected wound"). | 28 days following inititial treatment
Durability of wound closure (i.e., status of wound at one month following determination of "healed"). | 90 days following initial treatment
Serial wound punch biopsies for quantitative bacterial cultures, bacterial 16sRNA, and molecular analysis of 185 relevant wound healing genes. | 28 days following intitial treatment
Serum from venous blood and Vacuum Assisted Wound Closure Device (VAWCD) effluent for biomarkers, C-reactive protein, and cortisol levels. | 28 days following initial treatment
Mean wound surface area, circumference, depth and estimated volumes over time, ESWT group versus control group, as determined by CDM planimetry surface measurements. | 90 days following initial treatment
Length of hospital stay and number of surgical procedures for the extremity wound selected for study | 90 days following initial treatment
Assessment of relative burden of disease (trauma) between treatment groups by comparing mean values of the eight standard scales of the Medical Outcome Study 36-Item Short Form Health Survey (SF-36). | 90 days following intitial treatment

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Stojadinovic, MD, Principal Investigator — Walter Reed Army Medical Center
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Wang CJ. An overview of shock wave therapy in musculoskeletal disorders. Chang Gung Med J. 2003 Apr;26(4):220-32. PMID 12846521
- [Background] Wang CJ, Chen HS, Chen CE, Yang KD. Treatment of nonunions of long bone fractures with shock waves. Clin Orthop Relat Res. 2001 Jun;(387):95-101. doi: 10.1097/00003086-200106000-00013. PMID 11400901
- [Background] Schaden W, Fischer A, Sailler A. Extracorporeal shock wave therapy of nonunion or delayed osseous union. Clin Orthop Relat Res. 2001 Jun;(387):90-4. doi: 10.1097/00003086-200106000-00012. PMID 11400900
- [Background] Ludwig J, Lauber S, Lauber HJ, Dreisilker U, Raedel R, Hotzinger H. High-energy shock wave treatment of femoral head necrosis in adults. Clin Orthop Relat Res. 2001 Jun;(387):119-26. doi: 10.1097/00003086-200106000-00016. PMID 11400872
- [Background] Meirer R, Kamelger FS, Huemer GM, Wanner S, Piza-Katzer H. Extracorporal shock wave may enhance skin flap survival in an animal model. Br J Plast Surg. 2005 Jan;58(1):53-7. doi: 10.1016/j.bjps.2004.04.027. PMID 15629167
- [Background] Haupt G, Chvapil M. Effect of shock waves on the healing of partial-thickness wounds in piglets. J Surg Res. 1990 Jul;49(1):45-8. doi: 10.1016/0022-4804(90)90109-f. PMID 2359293
- [Background] Ludwig J, Lauber S, Lauber J, Hotzinger H. [Shockwave treatment of femur head necrosis in the adult]. Z Orthop Ihre Grenzgeb. 1999 Jul-Aug;137(4):Oa2-5. No abstract available. German. PMID 11051007
- [Background] Lauber S. [High energy extracorporeal shockwave therapy in femur head necrosis]. Z Orthop Ihre Grenzgeb. 2000 Sep-Oct;138(5):Oa3-4. No abstract available. German. PMID 11084728
- [Background] Gerdesmeyer L, von Eiff C, Horn C, Henne M, Roessner M, Diehl P, Gollwitzer H. Antibacterial effects of extracorporeal shock waves. Ultrasound Med Biol. 2005 Jan;31(1):115-9. doi: 10.1016/j.ultrasmedbio.2004.08.022. PMID 15653238